CLINICAL TRIAL: NCT06548503
Title: Assumption of Sylimarin, Pyrroloquinoline, Quinone Sodium Salt and Myricetin: Effects on Alcohol Levels and Markers of Oxidative Stress
Brief Title: Sylimarin, Pyrroloquinoline, Quinone Sodium Salt and Myricetin Assumption Effects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Gerardo Bosco, Associate Professor, University of Padova
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: SiPiMi2123
Record Dates: First submitted 2024-08-06; First posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Oxidative Stress; Alcohol Drinking
Keywords: oxidative stress; alcohol
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Intervention Model Description: Two groups, one with placebo, one with the Si.Pi.Mi product
Who Masked: Participant, Care Provider, Investigator
Masking Description: same taste, same case, just a letter on the external case.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Subject assumed the Si.Pi.Mi product as detailed in the protocol
  Interventions: Dietary Supplement: Si.Pi.Mi product
- Placebo (Placebo Comparator): Subjects assumed the placebo as detailed in the protocol
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Si.Pi.Mi product — Assumption of the product as detailed in the protocol
  Arms: Intervention
Other: Placebo — Assumption of placebo
  Arms: Placebo

SUMMARY:
Alcohol abuse is one of the most common causes of mortality worldwide, also associated with increased oxidative stress and end-organ damage in chronic assumption.

This study intend to evaluate the effect of the intake of a product contain silymarin, pyrroloquinoline quinone sodium salt, and myricetin (conventionally for this project Si.Pi.Mi.) on alcohol, ethyl glucuronide (EtG) and markers of oxidative stress levels on regular wine assumption over a predefined time period.

DETAILED DESCRIPTION:
The included subjects,will be randomized in a controlled, single-blinded trial to evaluate the intake of a product containing silymarin, pyrroloquinoline quinone sodium salt, and myricetin (conventionally for this project Si.Pi.Mi.) on alcohol levels and markers of oxidative stress.

Inclusion criteria:

* age between 18 and 35 years;
* no history of alcohol abuse or other substances.
* Caucasian ethnicity.
* no smoker;
* good health condition, no autoimmune, endocrine, infectious, cardiac, renal, hepatic or metabolic diseases;
* no pregnancy or lactation condition. Subjects will be asked to avoid the use of aspirin, paracetamol, or other anti-inflammatory drugs in the 7 days before and during the experiment and the assumption of caffeine in the 12 hours before the test. Furthermore, volunteers will be asked to avoid any alcoholic intake in the 7 days before and during the experiment except the one intended for the experiment.

All subjects will sign a consent after receiving proper information about the risks and benefits of this study.

Anthropometric data (height, weight, age) will be tracked at the beginning. Venous blood samples will be drawn for standardized clinical hematological analyses such as: mean cell volume (MCV), hepatic function including aspartate transferase (AST), alanine transferase (ALT), γ-glutamyltransferase (γ GT), total and fractionated bilirubin.

Experimental protocol

After inclusion, blind randomization using an electronic number generator will be performed into the following two groups:

A) placebo (sham-control) group. B) Si.Pi.Mi group. Subject and experimenters will be blinded to the group assignation.

2.2.1. Treatment and placebo Si.Pi.Mi. group will be supplemented with a commercial complex (AGfit3, Alchimia Innovazione srl, Padova, Italy). AGfit3, contains active agents coming from two plants: Silymarin and Myrica Cerifera, traditionally used for treating the liver, combined with the sodium salt of Bio-PQQ pyrroloquinoline quinone. AGfit3 is added to an aqueous solution of orange granular, freeze-dried orange, citric acid, sucrose. Placebo adopted is instead an aqueous solution of ascorbic acid (1 g), orange granular, freeze-dried orange, citric acid, sucrose.

In this experiment, all subjects will be asked to drink a glass (150 ml) of Cabernet red wine (Cantine Ca' Lustra Zanovello, Cinto Euganeo, PD, Italia) with an alcohol content of 12.5 ± 0.5%, corresponding to 14,81 - 15,40 g of ethanol according to a drink average dose as per current literature.

Biological samples will be collected, and measurements carried out as follows:

* Day 0: baseline before the experiment. Blood, saliva and urine samples collected (basal measures).
* Day 1: to evaluate acute wine intake, blood samples will be drawn 60, 120 and 240 min after drinking (150 mL of red wine) to establish ethanol metabolism curve. Placebo or Si.Pi.Mi. will be taken after the wine dose. Saliva will be collected 120 and 240 min after drinking while urine after 240 min.
* Day 2-6: long term intake - volunteers will drink one wine glass at lunch and another one at dinner (300 mL/die, corresponding to 30g ethanol/die approximately); they will assume the wine dose at the beginning of the meal, and then continue the diet with a balanced daily menu according to individual energy needs. They will then take placebo or Si.Pi.Mi. after the meal, depending on the group. Saliva will be collected in the morning.
* Day 7: biological samples will be collected in the same way as day 1 up to the end of the study.

Blood, saliva and urine samples After enrollment, for each subject, in the morning before breakfast, venous blood samples (about 5 mL) will be drowned in EDTA and LH tubes (Vacuette tube, Greiner bio-one, Kremsmünster, Austria), blood samples centrifugated (Hettich® MIKRO 200R centrifuge) for 10 min to separate plasma and red blood cells (RBC). Multiple aliquots then will be immediately frozen and stored at -80 °C. Plasma samples will be collected to determine blood ethanol, ROS, TAC, and Co Q10 levels. Saliva samples will be collected to determine ROS and TAC, while urine samples to determine Ethyl Glucuronoide (ETG), lipid peroxidation (8-iso-PGF2α) and NO metabolites (NOx), creatinine, neopterin, and uric acid concentration. Aminothiols' redox status will be evaluated by an RBC analysis.

Biomarker analysis

* Blood Alcohol Level Blood ethanol level will be determined using an Agilent 7820 A series GC instrument and HP-Innowax (30 m × 0.25 mm × 0.25 μm) capillary column, with Helium (flow = 1.5 mL/min) as carrier gas. The injector, the column and the detector will be maintained at 250 °C, 40 °C and 250 °C, respectively. The analysis will be carried out by isothermal elution. n-Propanol will be used as internal standard. Nitrogen, hydrogen and air will be used as gas for FID detector at 25, 40 and 400 mL/min, respectively.
* Urine Ethyl Glucuronoide (ETG) ETG is a metabolic product of ethylic alchool coming from the reaction of ethanol and acid glucuronic. ETG will be determined in urine samples using a commercial enzymatic immunoassay (quantILAB® n° W1510011723) according to manufacturer's instructions. All measures will be assessed in duplicate. The inter-assay coefficient of variation will be checked to fall in the range indicated by the manufacturer.
* Plasma ROS production An X-band electron paramagnetic resonance spectroscopy instrument (EPR, 9.3 GHz) (E-Scan, Bruker Co., Billerica, MA, USA) will be used to detect ROS production in plasma and saliva samples. Briefly, spin probe CMH (1-hydroxy-3-methoxy-carbonyl-2,2,5,5-tetramethylpyrrolidine) will be used for ROS de-termination while a stable radical CP (3-carboxy2,2,5,5-tetramethyl1-1-pyrrolidi-nyloxy) will be adopted as an external reference to convert ROS recorded data into absolute quantitative levels (µmol*min-1).
* Total Antioxidant Capacity (TAC) The 6-hydroxy-2,5,7,8-tetramethylchroman-2-carboxylic acid (Trolox-) equivalent antioxidant capacity assay, a widely used kit-based commercial method (Cayman Chemical, Ann Arbor, MI, USA, Item No. 709001), will be used as previously described [22, 24]. Briefly, 10 μL of plasma and/or saliva will be added in duplicate to 10 μL of metmyoglobin and then 150 μL of the chromogen solution; reactions will be started by the addition of 40 μL of hydrogen peroxide. Reaction mixtures will be incubated for 3 min at room temperature, then the absorbance signal at 750 nm will be determined by an Infinite M200 microplate reader spectrophotometer (Tecan, Austria). TAC will be expressed as trolox equivalent antioxidant capacity concentration (mM).
* 8-Isoprostane (8-iso-PGF2α) Lipid peroxidation will be assessed in urine samples using an immunoassay of 8-isoprostane concentration (Cayman Chemical, Ann Arbor, MI, USA, Item No. 516351). Samples and standard will be read in duplicate at a wavelength of 512 nm. Results will be normalized by urine creatinine values
* NO Metabolites NO derivatives, nitrate and nitrite (NO2 + NO3 = NOx), will be measured in urine samples by a colorimetric method based on the Griess reaction, using a commercial kit (Cayman Chemical, Ann Arbor, MI, USA; Item No. 780001). Samples will be read at 545 nm, and the concentration assessed by a standard curve.
* Co Q10 coenzyme CoQ10 plasma levels will be quantified using Human Coenzyme Q10 Elisa Kit (EKC33185, Biomatik, Ontario, Canada), following the manufacturer's instructions. Briefly, assay employs the competitive inhibition enzyme immunoassay technique; the microtiter plate provided in this kit has been pre-coated with CoQ10. Standards or plasma samples are added to the appropriate microtiter plate wells with Horseradish Peroxidase (HRP) conjugated antibody preparation specific for CoQ10. The competitive inhibition reaction is launched between with pre-coated CoQ10 and CoQ10 in samples. Samples will be read at 450 nm, and the concentration was assessed by a standard curve.
* Thiols measurement Total (tot) and reduced (red) aminothiols (Cys=cysteine, and GSH = glutathione) will be measured in erythrocytes (RBC). Thiol separation will be performed at room temperature by isocratic high-pressure liquid chromatography (HPLC) analysis on a Discovery C-18 column (250 × 4.6 mm I.D, Supelco, Sigma-Aldrich, St. Louis, MOS, USA), eluted with a solution of 0.1 M acetate buffer, pH 4.0: methanol, 81:19 (v/v), at a flow rate of 1 mL/min. Fluorescence intensities will be measured with an excitation wavelength at 390 nm and an emission wavelength at 510 nm, using a fluorescence spectrophotometer (Jasco, Japan). A standard calibration curve will be used.
* Creatinine, neopterin, and uric acid Urinary creatinine, neopterin, and uric acid concentrations will be measured in urine by isocratic high-pressure liquid chromatography (HPLC). The calibration curves will be linear over the range of 0.125-1 μmol/L, 0.625-20 mmol/L, and 1.25-10 mmol/L for neopterin, uric acid, and creatinine levels, respectively. Inter-assay and intra-assay coefficients of variation will be set at < 5%.
* Statistic analysis Kolmogorov-Smirnov test will be implemented to assess whether each variable followed a normal distribution, and descriptive statistics will be calculated. Two-way ANOVA with factors "type product" (Active vs Placebo) and "time" (1°day vs 7°day) will be applied. Then the one-way ANOVA will be applied to compare the trend values between the two groups. Tukey's honest tests will be used for post-hoc analysis. Probability levels of <0.05 will be considered significant. Also, the correlation between the investigated variables will be assessed using Spearman correlation coefficients. ROS production was considered as the primary outcome (no other parameters were taken into account), and prospective calculations of power to determine the sample size were made using G power software (GPower 3.1). At 80% power, the sample size-calculated in preliminary studies - has been set at eleven/ thirteen subjects.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 35 years;
* no history of alcohol abuse or other substances.
* Caucasian ethnicity.
* no smoker;
* good health condition, no autoimmune, endocrine, infectious, cardiac, renal, hepatic or metabolic diseases;
* no pregnancy or lactation condition.

Exclusion Criteria:

* pregnancy
* age falling outside limits
* smoke
* any disease

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Change in Reactive oxygen species production | Blood and Saliva: Day 0 (baseline); Day 1 and 7: 60, 120 and 240 min after drinking 150 mL of red wine + SiPiMi or placebo. On saliva alone: Day 2, Day 3, Day 4, Day 5, Day 6, in the morning.
  Reactive oxygen species production on blood and saliva (μmol/min) (by paramagnetic resonance)
Change in Total Antioxidant Capacity | Blood and Saliva: Day 0 (baseline); Day 1 and 7: 60, 120 and 240 min after drinking 150 mL of red wine + SiPiMi or placebo. On saliva alone: Day 2, Day 3, Day 4, Day 5, Day 6, in the morning.
  Total antioxidant capacity on blood and saliva (by paramagnetic resonance) (mM)
Change in lipid peroxidation markers | Day 1 and 7: at 0 and 240 min after drinking 150 mL of red wine + SiPiMi or placebo.
  Lipid peroxidation assessed by measuring 8-isoprostane and 8-OH deoxyguanosine concentration (by competitive immunoassay) (pg mg-1 creatinine)
Change in nitrite and nitrate (NO2 and NO3) concentration | Day 1 and 7: at 0 and 240 min after drinking 150 mL of red wine + SiPiMi or placebo.
  nitrite and nitrate (NO2 and NO3) concentration on urine (by colorimetry based on the Griess reaction (μM)
Change in Co Q10 coenzyme levels | Day 1 and 7: at 0 and 240 min after drinking 150 mL of red wine + SiPiMi or placebo.
  CoQ10 levels on blood (by competitive inhibition enzyme immunoassay) (μg/mL)
Change in aminothiols levels | Day 1 and 7: 0, 60, 120 and 240 min after drinking 150 mL of red wine + SiPiMi or placebo.
  total (tot) and reduced (red) aminothiols on blood (by fluorescence spectroscopy) (μmol L-1)
Change in Renal damage markers | Day 1 and 7: at 0 and 240 min after drinking 150 mL of red wine + SiPiMi or placebo.
  Renal damage by measuring on urine: creatinine (g-L-1), neopterin (μmol·mol-1 creatinine), and uric acid levels (mg/dl), (by isocratic high-pressure liquid chromatography)
Change in Blood Alcohol Levels | Day 1 and 7: 60, 120 and 240 min after drinking 150 mL of red wine + SiPiMi or placebo.
  Measurement of blood alcohol levels (g/L) (by isothermal elution)
Change in Urine Ethyl Glucuronoide | Day 1 and 7: at 0 and 240 min after drinking 150 mL of red wine + SiPiMi or placebo.
  Urine Ethyl Glucuronoide measurement on urine (ng/mL) (by enzymatic immunoassay)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Biomedical Sciences, Padua, Italy

IPD SHARING:
Plan to Share IPD: No
No sharing due to privacy reasons

REFERENCES:
- [Derived] Bosco G, Vezzoli A, Brizzolari A, Paganini M, Giacon TA, Savini F, Gussoni M, Montorsi M, Dellanoce C, Mrakic-Sposta S. Consumption of Sylimarin, Pyrroloquinoline Quinone Sodium Salt and Myricetin: Effects on Alcohol Levels and Markers of Oxidative Stress-A Pilot Study. Nutrients. 2024 Sep 3;16(17):2965. doi: 10.3390/nu16172965. PMID 39275279